CLINICAL TRIAL: NCT02396368
Title: A Phase I/Ib Study of Radium-223 in Combination With Tasquinimod in Bone-only Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of Radium-223 in Combination With Tasquinimod in Bone-only Metastatic Castration-Resistant Prostate Cancer
Acronym: Radium-223
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase III study results for the drug Tesquinimod were not promising so it was a drug development decision to stop using the drug
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1513; IRB00058873 (Other: JHMIRB)
Record Dates: First submitted 2015-02-25; First posted 2015-03-24 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer; Bone-only Metastatic Castration-Resistant Prostate Cancer (CRPC)
Keywords: Prostate cancer; Bone metastatic Castration-Resistant Prostate Cancer; Radium 223; Tasquinimod
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tasquinimod; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radium 223 and Tasquinimod (Experimental): During dose level 1, tasquinimod will start at 0.25mg/day orally with a goal of 0.5mg/day. Dose level 2 will start at 0.25mg/day with a goal of 1mg/day.
  Radium-223 will be administered per FDA-approved dosing (six IV injections at a dose of 50kBq/kg of body weight, administered every 4 weeks).
  Interventions: Drug: Tasquinimod; Radiation: Radium 223

INTERVENTIONS:
Drug: Tasquinimod — Tasquinimod is a quinoline-3-carboxamide analog that has demonstrated significant improvements in progression-free survival and overall survival in men with CRPC in a phase II trial.Tasquinimod will be administered at three dose levels (dose levels 1, 2, and -1). During dose level 1, tasquinimod will start at 0.25mg/day orally with a goal of 0.5mg/day. Dose level 2 will start at 0.25mg/day with a goal of 1mg/day. Dose level -1 will be 0.25mg/day without dose titration.
Radiation: Radium 223 — Radium Ra 223 dichloride, an alpha particle-emitting pharmaceutical, is a radiotherapeutic drug. Radium 223 is supplied as a clear, colorless, isotonic, and sterile solution to be administered intravenously with pH between 6 and 8. Each milliliter of solution contains 1,000 kBq radium-223 dichloride (27 microcurie), corresponding to 0.53 ng radium-223, at the reference date. Radium is present in the solution as a free divalent cation.Radium-223 will be administered per FDA-approved dosing (six IV injections at a dose of 50kBq/kg of body weight, administered every 4 weeks).

SUMMARY:
This is a Phase I/Ib study of Radium-223 in combination with Tasquinimod for patients with bone metastases from castration-resistant prostate cancer (CRPC).

The investigators propose to determine the spectrum of tolerability of the combination of tasquinimod and radium-223 and determine a dose for a subsequent randomized phase II study (first cohort) and the proportion of men with bone-specific alkaline phosphatase response (second cohort).

DETAILED DESCRIPTION:
This is a study of Radium-223 in combination with Tasquinimod. The target population is patients with bone metastases from castration-resistant prostate cancer intended for treatment with radium-223.

After baseline assessment, all subjects will receive six cycles of Radium-223 separated by an interval of 28 days. Radium-223 will be administered per FDA-approved dosing (six IV injections at a dose of 50kBq/kg of body weight, administered every 4 weeks). The treatment maintenance dose of tasquinimod will be a maximum of 1 mg of tasquinimod taken once daily with water (~200 mL). The initial target dose of tasquinimod is 0.5mg/day. All subjects will be followed up for 12 months after start of study treatment.

The investigators propose a phase I/Ib trial of the addition of tasquinimod to FDA-approved doses of radium-223 in men with symptomatic bone-only metastatic CRPC. The investigators anticipate that given their distinct mechanisms of action and non-overlapping toxicity profiles that additive or synergistic toxicity would be minimal. The investigators hypothesize that adding tasquinimod to radium therapy may result in improved measures of efficacy including reduction in total alkaline phosphatase, time to first skeletal-related event and PSA and radiographic progression-free survival.

In the Phase I portion of dose-escalation scheme, the dose escalation will follow a 3+3 design with intra-patient dose-escalation from 0.25mg/day of tasquinimod to a goal dose of either 0.25mg (dose-level -1), 0.5mg (dose-level 1), or 1.0mg/day (dose-level 2) based on individual tolerability.

Upon identifying a recommended Phase II combination dose-level of Radium-223 and tasquinimod, the investigators will move to the Phase Ib portion and open an expanded cohort of up to 35 additional patients to achieve a total of 38 patients treated at the recommended phase II dose-level (including those from the dose-escalation phase).

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years at the time of signing the ICF
2. Histologically or cytologically confirmed adenocarcinoma of the prostate
3. Two or more bone metastases (hot spots) confirmed by bone scintigraphy within 8 weeks prior to study entry
4. Pain at baseline judged by the investigator to be related to bone metastases
5. Known castration-resistant disease, defined according to PCWG2 criteria as:

   * Castrate serum testosterone level: ≤50 ng/dL (≤1.7 nmol/L)
   * Subjects who have failed initial hormonal therapy, either by orchiectomy or by using a GnRH agonist in combination with an anti-androgen, must first progress through antiandrogen withdrawal prior to being eligible. The minimum timeframe to document failure of anti-androgen withdrawal will be four weeks
   * Progressive disease based on PSA and/or radiographic criteria:Serum PSA progression defined as two consecutive increases in PSA over a previous reference value within 6 months of first study treatment, each measurement at least one week apart. Serum PSA at screening ≥ 2 ng/mL, Or Radiographic disease progression based on documented bone lesions by the appearance of two or more new lesions by bone scintigraphy
6. Karnofsky Performance Status (KPS): ≥70% within 14 days before start of study treatment (ECOG ≤1)
7. Life expectancy: at least 6 months
8. Laboratory requirements:

   * White Blood Cell (WBC) count ≥ 3 x 109/L
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x109/L
   * Hemoglobin ≥10.0 g/dL
   * Total bilirubin ≤ 1.5 x ULN
   * AST and ALT ≤ 3 x ULN
   * Creatinine ≤ 1.5 x ULN
9. If sexually active with partner of childbearing potential, patient will agree to use adequate contraceptive methods (barrier contraceptive with spermicide or vasectomy) while on study drug. The adequate contraceptive method should be continued for 6 months after the last dose of radium-223 or 14 days after the last dose of tasquinimod, whichever comes later.
10. No evidence (within 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin).
11. Able to swallow and retain oral medication.
12. The subject is willing and able to comply with the protocol, and agrees to return to the hospital for follow-up visits and examination
13. The subject has been fully informed about the study and has signed the informed consent form and, where appropriate, HIPAA authorization for release of personal health information

Exclusion Criteria:

1. Has received an investigational therapeutic drug within the last 4 weeks prior to start of study treatment, or is scheduled to receive one during the treatment period.
2. Has received external radiotherapy within the last 4 weeks prior to start of study treatment.
3. Previous therapy with antiandrogens within 4 weeks (within 6 weeks for bicalutamide eg, Casodex®).
4. Concurrent use of other anticancer agents or treatments, with the following exceptions:

   * Ongoing treatment with LHRH agonists or antagonists, denosumab (Prolia) or bisphosphonate (eg, zoledronic acid) is allowed. Ongoing treatment should be kept at a stable schedule; however, if medically required, a change of dose, compound, or both is allowed.
5. Any treatment modalities involving major surgery within 4 weeks prior to the start of study treatment.
6. Has received prior hemibody external radiotherapy.
7. Has received systemic radiotherapy (e.g. samarium, strontium etc.) for the treatment of bone metastases.
8. Has received blood transfusion or erythropoietin (EPO) within the last 4 weeks prior to start of study treatment.
9. Has received prior treatment with Radium-223.
10. Malignant lymphadenopathy exceeding 3 cm in short-axis diameter.
11. Symptomatic nodal disease, i.e. scrotal, penile or leg edema.
12. Visceral metastases from CRPC (>2 lung and/or liver metastases [size ≥2cm]), as assessed by CT scan or MRI of the chest/abdomen/pelvis within the last 8 weeks prior to start of study treatment.
13. Uncontrolled loco-regional disease.
14. Other primary tumor (other than CRPC) including hematological malignancy present within the last 5 years (except non-melanoma skin cancer or low-grade superficial bladder cancer).
15. Ongoing treatment with warfarin unless the international normalized ratio is well controlled and below 4. Treatment with other anticoagulants is allowed.
16. Maintenance treatment with corticosteroids corresponding to a prednisolone or prednisone dose above 10 mg/day. The dose must have been stable for at least 5 days.
17. Systemic exposure to ketoconazole or other strong CYP3A4 isozyme inhibitors or inducers (Appendix A) within 14 days prior to the start of study treatment. Systemic exposure to amiodarone is not allowed within 1 year prior to the start of study treatment.
18. Ongoing treatment with sensitive CYP1A2 substrate or CYP1A2 substrate with narrow therapeutic range (Appendix A) at the start of study treatment.
19. Ongoing treatment with CYP3A4 substrate with narrow therapeutic range (Appendix A) at the start of study treatment.
20. Has imminent or established spinal cord compression based on clinical findings and/or MRI.
21. Any other serious illness or medical condition that would, in the opinion of the investigator, make this protocol unreasonably hazardous, including, but not limited to:

    * Any uncontrolled infection
    * Cardiac failure NYHA (New York Heart Association) III or IV
    * Crohn's disease or ulcerative colitis
    * Bone marrow dysplasia
    * Known allergy to any of the compounds under investigation
    * Unmanageable fecal incontinence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Safety of combining Radium-223 with tasquinimod | Up to 18 months
  Safety of combining Radium-223 with tasquinimod will be assessed by the incidence and severity of toxicities (adverse events and serious adverse events).

SECONDARY OUTCOMES:
Bone-ALP response | Up to 18 months
  Bone-specific alkaline phosphatase (serum bone markers) response will be described as percentage of change from baseline to 6 months or earlier for those who discontinue study therapy
Time to radiographic or clinical progression or death, whichever comes first (progression free survival; PFS). | Up to 18 months
  Time to radiographic or clinical progression or death, whichever comes first (progression free survival; PFS). Based on RECIST version 1.1 and Prostate Cancer Working Group 2 (PCWG2) definitions including:
  1. Progression of soft tissue lesions according to RECIST 1.1
  2. Progression of bone lesions detected with bone scan according to PCWG2 criteria
  3. Radiologically-confirmed spinal cord compression or pathological fracture due to malignant progression
  4. Either of: time to first symptomatic SRE or symptomatic progression.
Time to first symptomatic SRE | Up to 18 months
  Time to first symptomatic SRE (defined as first use of XRT to relieve skeletal symptoms, new pathologic vertebral or nonvertebral bone fractures, spinal cord compression, or tumor -related orthopedic surgical intervention).
Proportion of patients without symptomatic progression at 6 months | 6 months
  To determine proportion of patients without symptomatic progression at 6 months, defined as any one or more of:
  1. Regular consumption of narcotic analgesics (single IV dose or >10 of 14 days of oral narcotic use)
  2. Requirement for radiation therapy for control of tumor-related pain
  3. VAS pain rating of >4 due to cancer pain on two consecutive ratings
Median change in the bone scan index (BSI) within patients at 12 weeks compared to baseline bone scan. | 12 weeks
PSA decline will be reported on all patients | 12 weeks
  The percentage of change in PSA from baseline to 12 weeks.
PSA progression (PSA progression free survival; PSA-PFS) | Up to 18 months
  PSA progression (PSA progression free survival; PSA-PFS) will be defined per the PCWG2 guidelines
  1. For those subjects showing an initial decline in PSA from baseline, is defined as an increase in PSA that is ≥25% and ≥2 ng/mL above the nadir, and which is confirmed by a second value 3 or more weeks later (i.e., a confirmed rising trend).
  2. For those subjects with no decline in PSA from baseline, is defined as an increase in PSA that is ≥25% and ≥2 ng/mL after 12 weeks.
Time to death after start of study treatment months | Up to 18 months
  Time to death after start of study treatment (overall survival; OS)
Changes in bone markers | Up to 18 months
  Changes in other bone markers:
  1. Serum C-telopeptide(uCTX-1)
  2. N-terminal propeptide of procollagen type 1 (P1NP)

OTHER OUTCOMES:
Radium-223 micro-scale dosimetry in bone tissue | Up to 18 months
  Radium-223 micro-scale dosimetry in bone tissue using bone biopsy material before and after treatment at 3 time points.
The spatial distribution of Ra-223 in the patient's skeleton | Up to 18 months
  Longitudinal whole-body planar gamma camera imaging will provide information on how tasquinimod impacts the overall skeletal distribution and uptake of Ra-223.
The whole organ-level dosimetry of Ra-223 in the the patient's skeleton | Up to 18 months
  Longitudinal whole-body planar gamma camera imaging will provide information on how tasquinimod impacts on the organ-level dosimetry and uptake of Ra-223.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Eisenberger, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States